CLINICAL TRIAL: NCT01599936
Title: Open Label, Confirmatory, Controlled Clinical Study of Alacramyn® in Pediatric Patients With Scorpion Sting Envenomation
Brief Title: Open Label Clinical Trial of Anascorp® in Pediatric Patients With Scorpion Sting Envenomation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Bioclon S.A. de C.V. (Industry)
Collaborators: University of Arizona (Other); Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-02/06
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Scorpion Sting
Keywords: scorpion sting; envenomation; Anascorp
MeSH Terms: conditions — Scorpion Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anascorp (Experimental): Three vials of Anascorp® will be administered in a total volume of 50 mL, intravenous over not less than 10 minutes or as permitted by IV access
  Interventions: Biological: Anascorp

INTERVENTIONS:
Biological: Anascorp — 3 vials of Alacramyn reconstituted in 50 ml of normal saline as an IV infusion over 10 minutes.
  Other Names: Antivenin Centruroides (scorpion) equine immune F(ab')2

SUMMARY:
There is no FDA approved therapy for the treatment of scorpion envenomation. Centruroides scorpion envenomation produces a pattern of neurotoxicity with a spectrum of severity ranging from trivial to life threatening. Patients stung by Centruroides scorpions develop a clinical syndrome which may require sedation with benzodiazepines and observation for 6 to 28 hours of intensive care monitoring. A safe therapy is necessary to halt the progression of symptoms early in the clinical course while avoiding the clinical deterioration that can occur en route to a tertiary facility. Alacramyn® is anticipated to be safer and more effective than the present standard of care, midazolam, and faster-acting thus eliminating the need to transport most rural patients and reducing hospitalization time.

DETAILED DESCRIPTION:
The purpose of this open label, confirmatory, controlled clinical trial was to examine the safety and efficacy of Alacramyn® for treatment of patients envenomed by scorpion sting.

This study took place at San Carlos Indian Hospital in San Carlos, Arizona and in two pediatric Intensive care units in Tucson, Arizona.

Patients who arrived at the emergency department presenting with scorpion sting symptoms were evaluated for treatment with respect to the inclusion/exclusion criteria according to the study procedures. Only patients with clinically important systemic signs of scorpion sting envenomation were included in the study. Baseline measures included severity evaluation of the scorpion sting envenomation. The patient's vital signs, concomitant medication, medical history and demographic data were collected. Blood tests were done for haematology, chemistry, venom and anti-venom levels and urine test.

After informed consent and inclusion/exclusion criteria were obtained and verified, and the baseline measurements completed, three vials of Alacramyn® were administered. At the one hour assessment an additional vial of Alacramyn® was administered if important systemic signs of scorpion envenomation were present. The assessment was repeated at two hours and a final vial of Alacramyn® was administered if deemed necessary. Patient were discharged after the 4 hour assessment if symptoms were resolved. Prior to discharge repeat lab work, physical assessments, and vital signs were done. Those remaining for extended care underwent final study assessments at time of hospital discharge or at 24 hours after study drug infusion if hospitalization continued.

All patients who participated in the study were contacted 7 and 14 days after treatment, looking for symptoms suggestive of ongoing venom effect, delayed serum sickness, as well as for any other adverse event reported by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 6 months to 18 years of age
* Presenting for emergency care within 5 hours with clinically important signs of scorpion sting envenomation
* Signed written Informed Consent by parent or legal guardian
* No participation in a clinical drug trial within the last month or concomitantly

Exclusion Criteria:

* Allergy to horse serum
* Use within the past 24 hours of drugs expected to alter immune response
* Use of any antivenom within the last month or concomitantly
* Underlying medical condition that significantly alters immune response
* Concurrent medical condition involving a baseline neurological status mimicking envenomation
* Pregnant and nursing women

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2004-04; Primary Completion 2006-10 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Resolution of clinically important systemic signs of scorpion envenomation within four hours after Alacramyn administration. | Assessments conducted at 1, 2 and 4 hours post administration

SECONDARY OUTCOMES:
Demonstrate that venom blood levels will decrease within one hour after Alacramyn® treatment. | One hour

CONTACTS AND LOCATIONS:
Overall Officials: Walter Garcia Ubbelohde, MD, Study Director — Instituto Bioclon; Leslie V. Boyer, MD, Principal Investigator — VIPER Institute, University of Arizona; Alejandro Alagon, PhD, Study Chair — Universidad Nacional Autonoma de Mexico
Locations (3):
- United States (3):
  - San Carlos Indian Hospital, San Carlos, Arizona
  - Tucson Medical Center, Tucson, Arizona
  - University Medical Center, Tucson, Arizona

REFERENCES:
- [Background] Boyer LV, Theodorou AA, Berg RA, Mallie J; Arizona Envenomation Investigators; Chavez-Mendez A, Garcia-Ubbelohde W, Hardiman S, Alagon A. Antivenom for critically ill children with neurotoxicity from scorpion stings. N Engl J Med. 2009 May 14;360(20):2090-8. doi: 10.1056/NEJMoa0808455. PMID 19439743
- [Background] Likes K, Banner W Jr, Chavez M. Centruroides exilicauda envenomation in Arizona. West J Med. 1984 Nov;141(5):634-7. PMID 6516334
- [Background] Gibly R, Williams M, Walter FG, McNally J, Conroy C, Berg RA. Continuous intravenous midazolam infusion for Centruroides exilicauda scorpion envenomation. Ann Emerg Med. 1999 Nov;34(5):620-5. doi: 10.1016/s0196-0644(99)70164-2. PMID 10533010
- [Background] Berg RA, Tarantino MD. Envenomation by the scorpion Centruroides exilicauda (C sculpturatus): severe and unusual manifestations. Pediatrics. 1991 Jun;87(6):930-3. No abstract available. PMID 2034501
- [Background] LoVecchio F, Welch S, Klemens J, Curry SC, Thomas R. Incidence of immediate and delayed hypersensitivity to Centruroides antivenom. Ann Emerg Med. 1999 Nov;34(5):615-9. doi: 10.1016/s0196-0644(99)70176-9. PMID 10533009
- [Background] Curry SC, Vance MV, Ryan PJ, Kunkel DB, Northey WT. Envenomation by the scorpion Centruroides sculpturatus. J Toxicol Clin Toxicol. 1983-1984;21(4-5):417-49. doi: 10.3109/15563658308990433. PMID 6381751